CLINICAL TRIAL: NCT04452227
Title: A Two-stage Translation of the Chinese Version Menstrual Distress Questionnaire: a Physical, Psychological, and Behavior Study in Taiwan
Brief Title: A Two-stage Translation of the Chinese Version Menstrual Distress Questionnaire
Status: Completed | Type: Observational
Sponsor: China Medical University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CMUH108-REC3-052
Record Dates: First submitted 2020-06-21; First posted 2020-06-30 (Actual); Last update posted 2020-06-30 (Actual); Status verified 2020-06

CONDITIONS: Non-disease State
Keywords: Menstrual Distress Questionnaire, Two-Stage Translation
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- eumenorrheic healthy women: women with a regular menstrual cycle for three months, predictable, and a period between 24-38 days that lasts less than 8 days.
  Interventions: Other: questionnaire

INTERVENTIONS:
Other: questionnaire — Filling the menstrual distress questionnaire, short-form McGill pain questionnaire, present pain index, visual analog scale

SUMMARY:
This study attempted to do the two-stage design of the translation of the MDQC (Menstrual Distress Questionnaire Form C-Cycle) Chinese version, and to do the validity and reliability test.

DETAILED DESCRIPTION:
Premenstrual syndrome is defined as recurrent moderate physical, psychological, behavior symptoms that occur during the luteal phase of menses and resolve with menstruation. It affects 20 to 32 percent of premenopausal women.

A diagnosis of PMS consists of determining the timing of the symptoms in relation to menses, meaningful change between post- and premenstrual symptom severity, and a clinically significant severity of the symptoms. The ICD-10 requires only one distressing symptom for a diagnosis of PMS. The American College of Obstetricians and Gynecologists (ACOG) diagnosis is that it occurs 5 days before menses and remit within 4 days of onset of menses no recurrence at least until day 13 of the cycle. A differential diagnosis to distinguish PMS from other medical and psychiatric conditions is important for appropriate treatment. No hormone or laboratory test indicates a PMS diagnosis. The current diagnostic standard requires confirmation of subjective symptom reports by prospective daily diaries. The Menstrual Distress Questionnaire (MDQ) is a method for measuring perimenstrual symptoms. It is a 46-item self-report inventory for use in the assessment of physical or psychological symptoms that occur in the premenstrual, menstrual, or intermenstrual phases. There are two forms of the MDQ: form C (Cycle) and form T (Today). Form C of the MDQ is designed for screening. Women use this form to describe their symptoms and reactions during each of the three phases of their most recent menstrual cycle. It may be administered at any time during the cycle. Form T is designed for treatment evaluation, and research application.

This study attempted to do the two-stage design of the translation of the MDQ (Form C-Cycle). Previous studies have translated only 14 items of the MDQ (Form C - Cycle) and only done the internal reliability test. This study is expected to do a two-stage translation of the MDQ (Form C - Cycle) Chinese version, and to do the reliability and validity test.

ELIGIBILITY:
Inclusion Criteria:

1. A eumenorrheic healthy woman with a regular menstrual cycle for three months, predictable, and a period between 24-38 days that lasts less than 8 days.
2. No hormonal contraceptives have been used in the past six months.
3. No history of smoking, drinking or drug abuse.

Exclusion Criteria:

1. Women with systemic diseases, cardiovascular diseases, liver diseases, kidney diseases, diabetes or thyroid diseases.
2. Taking any medicine due to chronic disease
3. Women with mental illness

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy females aged 20-40 years with regular and predictable menstrual cycles, fluent in speaking, reading, and writing Chinese in Taiwan
Sampling Method: Probability Sample
Enrollment: 219 (Actual)
Dates: Start 2019-06-22 (Actual); Primary Completion 2019-06-22 (Actual); Study Completion 2019-12-24 (Actual)

PRIMARY OUTCOMES:
questionnaire data | up to 8 weeks
  Statistical analyses were conducted using IBM SPSS Statistics 24 for Windows (IBM Inc., Armonk, NY, USA)

CONTACTS AND LOCATIONS:
Overall Officials: Su Shan-Yu, M.D. Ph.D., Principal Investigator — China Medical University Hospital
Locations (1):
- CMUH, Taichung, Taiwan